CLINICAL TRIAL: NCT02295410
Title: The Effects of Home-Based Telemental Health for Rural Veterans With PTSD
Acronym: HBTMH
Status: Completed | Type: Observational
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Collaborators: AnthroTronix, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2013-03/JLS 0007
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Assessment, PTSD, Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Engaged in Home-Based CPT: Home-Based Telemental Health-Patients undergoing Home-Based CPT for PTSD
  Interventions: Behavioral: CPT
- Comparison: Treatment as Usual (TAU) Patients NOT receiving regular CPT or other evidence-based therapy for PTSD.

INTERVENTIONS:
Behavioral: CPT
  Other Names: Cognitive Processing Therapy
  Groups: Engaged in Home-Based CPT

SUMMARY:
The intent of this study is to assess whether cognitive functioning improves as Post-Traumatic Stress Disorder (PTSD) symptoms decrease as a step toward developing an objective measure of PTSD improvement. The study also evaluates the feasibility and effectiveness of home-based telemental health care (HBTMH) compared to usual care in the treatment of rural Veterans with posttraumatic stress disorder (PTSD). For this assessment-only study, the investigators plan to assess approximately 200 Veterans in total, of which 150 will be undergoing regular evidenced-based therapy (EBT) for PTSD, and 50 will be receiving other treatment as usual (TAU). The 150 veterans in the EBT group will be undergoing Cognitive Processing Therapy (CPT), Cognitive-Behavioral Couple Therapy (CBCT), Prolonged Exposure (PE), or Seeking Safety (SS) treatment for PTSD in clinic or via home-based telemental health (HBTMH). The study will also assess a comparison group of approximately 50 rural Veterans with PTSD diagnoses who are receiving treatment as usual (TAU) (neither EBT nor HBTMH). The HBTMH patients will be recruited from an Office of Rural Health (ORH) funded project to VA Pacific Island Health Care System (VAPIHCS), based at the National Center for PTSD (NCPTSD) and funded to offer 100 rural Veterans mental health treatment in their homes. This research protocol intends to assess rural veterans with PTSD who are being seen within this clinic versus those who have been referred for HBTMH yet who are ineligible for pragmatic purposes, with outcomes including feasibility, cost-effectiveness, and clinical effectiveness. The cognitive change will also be measured in patients with PTSD diagnoses receiving EBT PTSD treatment at VA clinics in the Pacific Islands.

DETAILED DESCRIPTION:
The Office of Rural Health has funded the VA Pacific Islands Healthcare System (VAPIHCS) to provide HBTMH for rural veterans diagnosed by a mental health provider as having PTSD. VAPIHCS serves an area about the size of the continental United States. Outside of Honolulu, there are few mental health specialists to serve Veterans with PTSD and common comorbid disorders, such as traumatic brain injury (TBI), pain, insomnia, and substance abuse. Moreover, many such Veterans have difficulty following-up for services at Community-Based Outpatient Clinics (CBOCs) due to psychological or physical limitations, transportation, work schedule, or stigma.

Cost is another reason to develop a HBTMH approach. Seventy percent of those who complete a course of Evidence Based Therapy (EBT) significantly improve their symptoms, with most no longer carrying the diagnosis following such treatments (Bradley, Greene, Russ, Dutra, & Westen, 2005). However those who lack access to EBTs, especially those with polytraumas, have a low chance of recovery (Elhers & Clark, 2008; Lyons & Keane, 1992). The lack of specialists in these regions means that the Veterans continue to suffer with PTSD and related disorders far longer than if specialized care were available. Sending experts to these areas is costly, and inefficient. The cost and difficulty for highly rural Veterans to travel for weekly appointments to a CBOC that lacks expertise in EBT for PTSD and treating Veterans with polytrauma has minimal value. Finally, the no-show rate for such Veterans can run well above 15%, whereas research with HBTMH has no-show rates of less than 4% (http://conference.avapl.org/pubs/2012%20Conference%20Presentations/HBTMH%20SOP_Shore_11-12-11%20copy.pdf)

To improve services for Veterans, the VA provides telehealth options at its CBOC locations in the Pacific Islands. Many patients live too far from the CBOC or prefer to receive mental health treatment in the comfort of their own homes. HBTMH technology, such as televideo sessions between a home-based patient and their mental healthcare provider, has been successfully implemented in the VA (e.g. throughout VISN 20 and VISN 7) and in the Department of Defense (DOD). VAPIHCS was funded by the ORH to provide evidence-based specialty treatment via HBTMH to rural Veterans with PTSD who would not otherwise have such treatment available to them. The clinical project is funded to provide up to 100 rural patients who were referred by their CBOC providers to this specialty clinic for HBTMH PTSD treatment. This VAPIHCS clinic provides evidence-based treatment to eligible veterans in their homes via televideo by clinicians currently based at the NCPTSD. Only ORH-funded VAPIHCS clinical staff will provide treatment to the PTSD patients who choose to and are eligible to receive the home-based telemental health. Veterans are eligible for this VAPIHCS-HBTMH clinic if they have been diagnosed with PTSD by a licensed mental health provider at a CBOC, or are referred by a CBOC (via clinical consult).

In order to initially evaluate the effectiveness of HBTMH, the current research study will evaluate veterans participating in the VAPIHCS-HBTMH clinic compared to Treatment as Usual (TAU - those who were referred to the clinic, however either refused to participate in this type of clinical care or were ineligible to be part of this clinic due to structural difficulties (no 4G in their area, can't type, lack of nearby emergency services, etc). Thus, this protocol is assessment only, and is separate from the treatment provided to the rural Veterans.

Currently, there are no standardized, objective assessments available for determining impairment and improvement of PTSD. The Defense Automated Neurobehavioral Assessment (DANA) is a clinical decision support tool developed for the Department of Defense (DoD) for field and clinic-based neurobehavioral functioning. This neurobehavioral assessment system was developed on the assumption that various risk factors (PTSD, Depression, Insomnia, anger, pain, etc.) lead to significantly slower and less accurate (throughput) performance on cognitive tests. The primary goal of DANA is to assist providers in determining level of functioning and to track recovery over time. An important purpose of this study is to collect longitudinal data from patients receiving EBT (both in clinics and through HBTMH) in order to assess whether cognitive functioning improves as PTSD symptoms decrease with treatment. This information will provide support for DANA's validity as an objective measure of PTSD impairment. The study also plans to determine the sensitivity and specificity of DANA neurocognitive measures in determining changes in cognitive functioning within PTSD patients engaged in EBT over time.

The proposed project aims to examine the effectiveness of an empirically based trauma-focused treatment intervention delivered via video conferencing to the home. This project aims to:

Objective 1: Examine the feasibility of HBTMH compared to treatment as usual.

Objective 2: Compare the effectiveness of HBTMH compared to treatment as usual.

Objective 3: Determine predictors of successful treatment outcomes (including treatment completion and clinically significant reduction in PTSD and related symptoms).

Objective 4: Determine the sensitivity and specificity of Defense Automated Neurobehavioral Assessment (DANA) neurocognitive measures in determining changes in psychological functioning within subjects over time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a referral to the HBTMH Clinic or VA clinic for PTSD treatment as well as:

  1. ability to use a keyboard
  2. the ability to demonstrate a thorough understanding of the study and willingness to participate
  3. comfort using a tablet device and the Internet, or willingness to learn
  4. have agreed to return the tablet and headset after the study (TAU and HBTMH-only)
  5. adequate (or corrected) vision and hearing
  6. ability to read and write at an 8th grade level or higher.

Exclusion Criteria:

1. clinical disqualification (current psychosis, active homicidal or suicidal intent or within the past six months)
2. significant cognitive impairment as determined by inability to sufficiently comprehend the study goals, risks and benefits.

   * To determine this, potential research participants will be asked to summarize the study as explained to them and as presented by the Study Fact Sheet/Consent Form as applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 Veterans with PTSD who have been referred by their CBOC to the HBTMH PTSD clinic or a VA Clinic will be enrolled in this research study. This sample size is based on the number of treatment subjects intended to be treated by the HBTMH clinic, the VA clinic, and the estimated numbers of subjects who will be ineligible or choose not to participate in the HBTMH treatment. This number should be sufficient given past effect size differences between HBTMH treatment and TAU (Cohen's d effect size averaging about 1.0). It will also allow us to measure changes in psychological and cognitive functioning within treatment subjects over time.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in PCL-M | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Posttraumatic Stress Disorder Checklist- Military (PCL-M) [repeated measure]

SECONDARY OUTCOMES:
Change in Simple Reaction Time Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of Reaction time speed and accuracy. [repeated measure]
Change in Procedural Reaction Time Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of Procedural Reaction time speed and accuracy. [repeated measure]
Go-No Go Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of IsFoe or IsNotFoe for speed and accuracy. [repeated measure]
Change in Code Substitution (Learning and Recall) Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of Code Substitution (Learning and Recall) for speed and accuracy. [repeated measure]
Change in Spacial Processing Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of Spacial Processing for speed and accuracy. [repeated measure]
Change in Matching to Sample Throughput | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Computerized Neurocognitive Test of Matching to Sample for speed and accuracy. [repeated measure]
Change in PHQ-9 | approximately 0, 4 and 8 weeks depending on the number of CPT sessions completed.
  Patient Health Questionnaire -9 for measuring depression [repeated measure]

CONTACTS AND LOCATIONS:
Overall Officials: James Spira, PhD, Principal Investigator — NPTSD
Locations (1):
- VA Pacific Island Health Care System, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Lathan C, Spira JL, Bleiberg J, Vice J, Tsao JW. Defense Automated Neurobehavioral Assessment (DANA)-psychometric properties of a new field-deployable neurocognitive assessment tool. Mil Med. 2013 Apr;178(4):365-71. doi: 10.7205/MILMED-D-12-00438. PMID 23707818
- [Background] Spira JL, Lathan CE, Bleiberg J, Tsao JW. The impact of multiple concussions on emotional distress, post-concussive symptoms, and neurocognitive functioning in active duty United States marines independent of combat exposure or emotional distress. J Neurotrauma. 2014 Nov 15;31(22):1823-34. doi: 10.1089/neu.2014.3363. Epub 2014 Oct 9. PMID 25003552